CLINICAL TRIAL: NCT04519437
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study Assessing the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of Repeated Subcutaneous Doses of Anti-Spike (S) SARS-CoV-2 Monoclonal Antibodies (REGN10933+REGN10987) in Adult Volunteers
Brief Title: Study Assessing the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of Repeated Subcutaneous Doses of Anti-Spike (S) SARS-CoV-2 Monoclonal Antibodies (REGN10933+REGN10987) in Adult Volunteers as Related to COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R10933-10987-HV-2093
Record Dates: First submitted 2020-07-24; First posted 2020-08-19 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Healthy; Chronic Stable Illness
Keywords: Coronavirus disease 2019 (COVID-19); Severe acute respiratory syndrome coronavirus 2 (SARS-COV-2)
MeSH Terms: conditions — COVID-19 | interventions — casirivimab and imdevimab drug combination; casirivimab; imdevimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- REGN10933+REGN10987 (Experimental)
  Interventions: Drug: REGN10933+REGN10987
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: REGN10933+REGN10987 — Administered subcutaneous (SC) every 4 weeks (Q4W)
  Other Names: REGN-COV2; Casirivimab; Imdevimab; REGEN-COV™; Ronapreve™
  Arms: REGN10933+REGN10987
Drug: Placebo — Administered subcutaneous (SC) every 4 weeks (Q4W)
  Arms: Placebo

SUMMARY:
The primary objectives are:

* To assess the occurrence of adverse events of special interest (AESIs) in participants treated with repeated subcutaneous (SC) doses of REGN10933+REGN10987 compared to placebo
* To assess the concentrations of REGN10933 and REGN10987 in serum over time after single and repeated SC administration

The secondary objectives are:

* To assess the safety and tolerability of repeated SC doses of REGN10933+REGN10987 compared to placebo
* To assess attainment of target concentrations of REGN10933 and REGN10987 in serum after single and repeated SC administration
* To assess the immunogenicity of REGN10933 and REGN10987

ELIGIBILITY:
Key Inclusion Criteria:

1. Is healthy or has chronic medical condition(s) that is stable and well controlled as per the opinion of the investigator and is not likely to require medical intervention through the end of study
2. Stable medication for co-morbid condition(s) for at least 6 months prior to screening
3. Willing and able to comply with study visits and study-related procedures, including compliance with site precautionary requirements related to SARS-CoV-2 infection and transmission

Key Exclusion Criteria:

1. Positive diagnostic test for SARS-CoV-2 infection ≤72 hours prior to randomization
2. Subject-reported clinical history of COVID-19 as determined by investigator
3. Subject-reported history of prior positive diagnostic test for SARS-CoV-2 infection
4. Active respiratory or non-respiratory symptoms suggestive or consistent with COVID-19
5. Medically attended acute illness, systemic antibiotics use, or hospitalization (ie, >24 hours) for any reason within 30 days prior to screening
6. Acute exacerbation of a chronic pulmonary condition (eg, chronic obstructive pulmonary disease [COPD], asthma exacerbations) in the past 6 months prior to screening
7. Received investigational or approved SARS-CoV-2 vaccine
8. Received investigational or approved passive antibodies for SARS-CoV-2 infection prophylaxis as defined in the protocol
9. Use of remdesivir, intravenous immunoglobulin (IVIG), or other anti-SARS viral agents within 2 months prior to screening

NOTE: Other protocol-defined Inclusion/ Exclusion criteria apply

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 974 (Actual)
Dates: Start 2020-07-26 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2021-11-22 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse event of special interests (AESIs) that occur within 4 days of study drug administration | Within 4 days postdose at Baseline
Incidence of adverse event of special interests (AESIs) that occur within 4 days of study drug administration | Within 4 days postdose at Day 29
Incidence of adverse event of special interests (AESIs) that occur within 4 days of study drug administration | Within 4 days postdose at Day 57
Incidence of adverse event of special interests (AESIs) that occur within 4 days of study drug administration | Within 4 days postdose at Day 85
Incidence of adverse event of special interests (AESIs) that occur within 4 days of study drug administration | Within 4 days postdose at Day 113
Incidence of adverse event of special interests (AESIs) that occur within 4 days of study drug administration | Within 4 days postdose at Day 141
Concentrations of REGN10933 in serum over time | Up to 52 weeks
Concentrations of REGN10987 in serum over time | Up to 52 weeks

SECONDARY OUTCOMES:
Proportion of participants with treatment-emergent adverse events (TEAEs) | Up to 52 weeks
Severity of TEAEs | Up to 52 weeks
Proportion of participants who achieve or exceed target concentration in serum of REGN10933 | Up to 52 weeks
Proportion of participants who achieve or exceed target concentration in serum of REGN10987 | Up to 52 weeks
Immunogenicity as measured by anti-drug antibodies (ADA) to REGN10933 | Up to 52 weeks
Immunogenicity as measured by anti-drug antibodies (ADA) to REGN10987 | Up to 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (7):
- United States (7):
  - Regeneron Study Site, Tempe, Arizona
  - Regeneron Study Site, Rogers, Arkansas
  - Regeneron Study Site, Sacramento, California
  - Regeneron Study Site, Miami, Florida
  - Regeneron Study Site, Lincoln, Nebraska
  - Regeneron Study Site, Dayton, Ohio
  - Regeneron Study Site, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual anonymized participant data will be considered for sharing once the indication has been approved by a regulatory body, if there is legal authority to share the data and there is not a reasonable likelihood of participant re-identification.
Access Criteria: Qualified researchers may request access to anonymized patient level data or aggregate study data when Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency [EMA], Pharmaceuticals and Medical Devices Agency [PMDA], etc) for the product and indication, has the legal authority to share the data, and has made the study results publicly available (eg, scientific publication, scientific conference, clinical trial registry).
URL: https://vivli.org

REFERENCES:
- [Derived] Hirsch C, Park YS, Piechotta V, Chai KL, Estcourt LJ, Monsef I, Salomon S, Wood EM, So-Osman C, McQuilten Z, Spinner CD, Malin JJ, Stegemann M, Skoetz N, Kreuzberger N. SARS-CoV-2-neutralising monoclonal antibodies to prevent COVID-19. Cochrane Database Syst Rev. 2022 Jun 17;6(6):CD014945. doi: 10.1002/14651858.CD014945.pub2. PMID 35713300
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343